CLINICAL TRIAL: NCT05931224
Title: A Randomized, Double-blind, Multi-center, Therapeutic Confirmatory, Phase 3 Trial To Evaluate the Efficacy and Safety of D064 and D702 Combination Therapy Versus D660 Monotherapy in Essential Hypertension Patients
Brief Title: Clinical Trial to Evaluate the Efficacy and Safety of D064 and D702 Combination Therapy
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Chong Kun Dang Pharmaceutical (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: A30_15HT2213
Record Dates: First submitted 2023-06-27; First posted 2023-07-05 (Actual); Last update posted 2024-06-04 (Actual); Status verified 2024-06

CONDITIONS: Essential Hypertension
MeSH Terms: conditions — Essential Hypertension | interventions — 2-(3,4-dimethoxyphenyl)-8-(4-hydroxy-3-methoxyphenyl)-6-methyl-2-isopropyl-6-azaoctanitrile

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental Group (Experimental)
  Interventions: Drug: D064, D702, placebo of D660
- Comparator Group (Experimental)
  Interventions: Drug: D660, placebo of D064, placebo of D702

INTERVENTIONS:
Drug: D064, D702, placebo of D660 — Experimental Group Subjects assigned to this group are treated with D064, D702, placebo of D660
  Other Names: D064, D702 are consisted of antihypertensive agent.
  Arms: Experimental Group
Drug: D660, placebo of D064, placebo of D702 — Experimental Group Subjects assigned to this group are treated with D660, placebo of D064, placebo of D702
  Other Names: D660 is consisted of antihypertensive agent.
  Arms: Comparator Group

SUMMARY:
Clinical Trial to Evaluate the Efficacy and Safety of D064 and D702 Combination Therapy

ELIGIBILITY:
Inclusion Criteria:

* Subjects who are 19 years old or older.
* Subjects who have voluntarily decided to participate in this clinical trial and signed ICF.

Exclusion Criteria:

1. Subjects with a history of secondary hypertension or suspected secondary hypertension
2. Subjects with hypersensitivity or history of clinical trial drugs and similar drugs
3. Subjects who are required to administer a combination of prohibited drugs specified in this plan during the clinical trial participation period
4. Subjects with a history of drug or alcohol abuse or suspected patient within 24 weeks as of the time of screening
5. Subjects who received other clinical trial drugs within 4 weeks of screening visit.
6. Pregnant women, lactating women, or Subjects who do not agree to use appropriate contraception during the clinical trial period and for two weeks after the end of administration of the last clinical trial drug
7. Subjects who are unable to participate in this clinical trial at the discretion of the investigator.

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 346 (Actual)
Dates: Start 2023-06-28 (Actual); Primary Completion 2024-05-13 (Actual); Study Completion 2024-05-13 (Actual)

PRIMARY OUTCOMES:
Change from baseline in MSSBP | 8 weeks after drug administrations
  MSSBP(Mean Sitting Systolic Blood Pressure)

CONTACTS AND LOCATIONS:
Overall Officials: Inho Chae, M.D, Ph.D, Principal Investigator — Seoul National University Bundang Hospital
Locations (1):
- Seoul National University Bundang Hospital, Seongnam, Bundang-gu, South Korea

IPD SHARING:
Plan to Share IPD: No